CLINICAL TRIAL: NCT04172285
Title: Effects of an Home-base Physical Activity Program for Counteracting Sarcopenia in Elderly: a Randomized-controlled Trial.
Brief Title: Physical Activity Program for Counteracting Sarcopenia
Acronym: EXERSARCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXERSARCO
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical activity group (Experimental)
  Interventions: Behavioral: Physical activity
- Physical activity and supplementation group (Experimental)
  Interventions: Dietary Supplement: Physical activity and supplementation
- Control group (Experimental)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Physical activity — Home-based physical activity program
  Arms: Physical activity group
Dietary Supplement: Physical activity and supplementation — Home-based physical activity program and amminoacid supplementation
  Arms: Physical activity and supplementation group
Other: Control — No intervention
  Arms: Control group

SUMMARY:
Sarcopenia is a pathophysiological process associated with aging and some metabolic conditions characterized by progressive muscle tissue loss, which may lead to loss of strangth and performance and increase risk of falls and fractures, physical disability and premature death. Therefore, it is necessary to identify personalized programs of physical activity and supplementation for elderly population in order to improve their physical functions, muscle strengh and body composition.

With the present project we aime to assess the effect of a feasible home-based exercise program coupled with food supplementation to improve muscle strength, muscle volume and muscle physical performance potentially associated with sarcopenia in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle.
* Cognitively intact.
* Autonomous walking.
* Acceptance of informed consent.

Exclusion Criteria:

* Body mass index lower than 18.5 and uppen than 40 kg/m2.
* History of cancer.
* Pacemaker user.
* History of epileptic episodes.
* Endocrine-metabolic, neurological, muscular and ortopedic pathologies that affect movement functions.
* Bone fractures that influence movement functions.
* Smoking.
* Surgical treatments in the prior 6 months.
* Use of antieptilectics, glucocorticoids, rhGH and testosterone.
* Hepatic and muscular pathologies

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Lower limb strength | Baseline and Week 24
  Assessed by chair stand test

SECONDARY OUTCOMES:
Body composition | Baseline and Week 24
  Assessed by Whole-body dual energy X-ray absorptiometry
Quantify thigh cross sectional area | Baseline and Week 24
  Assessed by Dixon magnetic resonance imaging
Maximum isometric force that a hand can squeeze | Baseline and Week 24
  Assessed by Hand Grip Strength test
Maximal Isometric Strength of Knee flexors and extensors | Baseline AND Week 24
  Assessed by a belt-stabilized dynamometer
Dynamic balance and gait deficits | Baseline and Week 24
  Assessed by mini-BESTest

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy